CLINICAL TRIAL: NCT05764382
Title: Remote Tai Ji for Low Back Pain: a Randomized Trial
Brief Title: Remote Tai Ji for Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Presbyterian Hospital (Other)
Collaborators: Center for Taiji and Qigong Studies & Wa-Qi.com (Unknown)
Responsible Party: Principal Investigator, Pravesh Gadjradj, Physician, Epidemiologist, New York Presbyterian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27012023
Record Dates: First submitted 2023-01-27; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: Tai Chi; Qigong
MeSH Terms: conditions — Low Back Pain | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T'ai Chi and Qigong Rehabilitation (Experimental)
  Interventions: Behavioral: T'ai Chi and Qigong Rehabilitation
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: T'ai Chi and Qigong Rehabilitation — T'ai chi/Qigong is a multidimensional (mind, body, and spirit integrative) and multimodal (strength, flexibility, balance, posture, and light to moderate aerobic) form of exercise that is safe for persons of all ages and physical abilities. The 12-week, twice-per-week t'ai chi and qigong gentle movement and meditation program proposed to be studied is adapted from the WaQi program, a curriculum developed by Master Yang Yang, PhD. Master Yang developed this course based on his own healing journey from severe back pain following a bike accident in 2014.
  Arms: T'ai Chi and Qigong Rehabilitation
Other: Usual care — Usual care as per primary care physican, physical therapist.
  Arms: Usual care

SUMMARY:
The purpose of the study is to examine the implementation strategy, in terms of feasibility and the possible benefits, of a free online Zoom t'ai chi and qigong gentle movement and meditation program to reduce back pain and to improve sleep and quality of life among those with chronic back pain. The primary objective of this study is to examine whether a safe and moderate online t'ai chi and qigong exercise program, offered without cost to individuals with chronic back pain, improves pain levels, sleep, and quality of life; The secondary objective is to explore whether improvements in pain levels are different among smokers and those with unhealthy BMI than among others.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Have experienced low back pain for the last 6 weeks or longer
* Understands written and spoken English
* Be willing to complete the initial survey and 3 additional ones emailed baseline and January 2023
* Be willing and able to provide consent to participate in the survey

Exclusion Criteria:

* pregnany
* previously has taken t'ai chi classes
* spine surgery within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Oswestry Disability Index 3 months after intervention | baseline, 3 months
  0 to 100 scale

SECONDARY OUTCOMES:
Change in visual analogue scale (VAS) for low back pain | baseline, 3 months
  0-100 scale
Change in VAS leg pain | baseline, 3 months
  0 to 100 scale
The "SF-36," Short Form Health Survey questionnaire | baseline, 3 months
9-Item Pittsburgh Sleep Quality Index | baseline, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, PhD, Study Director — Director Center for Taiji and Qigong Studies & Wa-Qi.com https://www.wa-qi.com
Locations (1):
- New York Presbytarian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided